CLINICAL TRIAL: NCT05398822
Title: The Role of TextRAd on Detection of Liver Metastasis in Rectal Cancer
Status: Completed | Type: Observational
Sponsor: East Suffolk and North Essex NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 19/109
Record Dates: First submitted 2022-05-26; First posted 2022-06-01 (Actual); Last update posted 2022-06-01 (Actual); Status verified 2022-05

CONDITIONS: Rectal Cancer
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: MRI — Texture analysis (TA) is a novel imaging biomarker that can assess heterogeneity in MRIs by measuring grey-level intensities distribution. This study hypothesizes that TA of MRI is an imaging biomarker that can predict local recurrence and distant metastasis.

SUMMARY:
This is a retrospective analysis of all patients diagnosed with LARC who received NCRT and had MRI scans between 2003-2014 at East Suffolk and North Essex NHS Foundation Trust. Region of interest was drawn around the tumor or its location on T2 MRI images. Six texture parameters were systematically extracted from Textural histograms of post-treatment scans. These parameters were examined to determine their ability to predict local recurrence and distant metastases through Kaplan-Meier survival curves and log-rank tests.

ELIGIBILITY:
Inclusion Criteria:

* All subjects must have MRI post-Chemotherapy treatment to detect the response to Neoadjuvant treatment and compare it to pre-treatment scans to easily determine if there were a posttreatment liver metastasis.
* Locally advanced rectal cancer (LARC) = MRI stage: T3/T4 and/or N1/N0.

Exclusion Criteria:

* Distant metastases.
* Synchronous tumour.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients diagnosed with locally advanced rectal cancer (LARC) includes neoadjuvant chemoradiotherapy (NCRT) followed by surgical resection
Sampling Method: Non-Probability Sample
Enrollment: 113 (Actual)
Dates: Start 2019-07-18 (Actual); Primary Completion 2021-07-18 (Actual); Study Completion 2021-07-18 (Actual)

PRIMARY OUTCOMES:
Local recurrence of rectal cancer | 120 months

CONTACTS AND LOCATIONS:
Locations (1):
- East Suffolk and North Essex NHS Foundation Trust, Ipswich, United Kingdom

IPD SHARING:
Plan to Share IPD: No